CLINICAL TRIAL: NCT01932866
Title: Impact of a Diabetes Risk Score on Lifestyle Education and Patient Adherence (IDEA Trial)
Brief Title: Impact of a Diabetes Risk Score on Lifestyle Education and Patient Adherence
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark True, MD, Program Director, Endocrinology Fellowship, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDEA Trial
Record Dates: First submitted 2013-08-21; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Pre-diabetes; Diabetes Risk Score; Motivation
Keywords: pre-diabetes; diabetes risk score; motivation; Air Force; Military; Lifestyle change
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control - diabetes risk score (Active Comparator): the participants in the control group did not receive their diabetes risk score at the beginning of the trial, but did receive their scores to include baseline at the 12 and 24 week points.
  Interventions: Other: diabetic risk score
- Intervention - diabetes risk score (Experimental): the subjects in the intervention arm received their diabetes risk scores at the beginning of the trial, 12 weeks and 24 weeks.
  Interventions: Other: diabetic risk score

INTERVENTIONS:
Other: diabetic risk score

SUMMARY:
The purpose of this randomized, controlled study is to evaluate whether the knowledge of a personalized diabetes risk score affects adherence to a 12-week diet and exercise lifestyle change program in prediabetic patients. The intervention group will receive diabetes risk score results at the beginning of the twelve weeks, and the control group will not receive these results. Both groups will review their baseline and 12-week diabetes risk score results at the conclusion of the program and will be followed for an additional twelve weeks. Attendance rates and changes in weight, BMI, abdominal circumference, blood pressure, HgA1c, fasting blood glucose, cholesterol, and diabetes risk score will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of all ethnic groups
* ≥30 -75 years of age
* Pre-diabetic defined as follows: fasting plasma glucose (FPG) 100-125mg/dL, HbA1c 5.7% to 6.4%.
* Body Mass Index ≥ 25 kg/m2
* Tricare beneficiary

Exclusion Criteria:

Diagnosis of type 1 or type 2 diabetes mellitus (defined as FPG ≥126 mg/dl on two different occasions or random blood sugar ≥200) If fasting glucose >= 126 only once, a second lab does not need to be arranged in an attempt to diagnose diabetes. It is acceptable for the patient to proceed in the trial. Also, Tethys lab results (e.g., fasting glucose and A1C) should not be used to make decisions about including or excluding patients in the trial. Only Air Force lab results should be used to make this determination.

* Active duty military members
* Patients with untreated hypothyroidism or previously diagnosed Cushing's syndrome
* Subjects previously treated with metformin or thiazolidinediones in the previous 12 months
* Psychological or physical disabilities deemed likely to interfere with participation in the study
* Patients currently using weight-loss medications or medications known to affect body weight (i.e. chronic corticosteroid use)
* Major medical conditions that prevent participation in the Group Lifestyle Balance Prevention Program (i.e. severe cardiovascular or cerebrovascular disease, severe renal or liver dysfunction, etc.)
* Concurrent participation in a different weight loss program
* Previous bariatric surgery
* Unwilling to agree with the study assignments or provide informed consent
* Participation in any other research project that would interfere with this protocol
* Unable to read and write English
* Pregnant or nursing patients
* Female patients unwilling to undergo a pregnancy test or report possible pregnancy promptly and unwilling to take precautions to avoid pregnancy if potentially fertile during the study course

Discontinuation Criteria:

* Consent is withdrawn
* Death occurs
* A woman becomes pregnant
* Severe impairment of manual dexterity, vision, or intellectual function
* They become lost to follow-up because of a move or transfer outside of the geographic area

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Attendance rates | 6 months
  Attendance rates (percentage of subjects attending the classes) of the two groups will be compared.
Change in weight | baseline, 12 weeks, 24 weeks
  change in weight from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in BMI | baseline, 12 weeks, 24 weeks
  change in BMI from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in abdominal circumference | baseline, 12 weeks, 24 weeks
  change in abdominal circumference from baseline to 12 weeks and 24 weeks will be compared between groups.

SECONDARY OUTCOMES:
Change in blood pressure | baseline, 12 weeks, 24 weeks
  change in blood pressure from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in HgA1c | baseline, 12 weeks, 24 weeks
  change in HgA1c from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in fasting blood glucose | baseline, 12 weeks, 24 weeks
  change in fasting blood glucose from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in cholesterol | baseline, 12 weeks, 24 weeks
  change in cholesterol from baseline to 12 weeks and 24 weeks will be compared between groups.
Change in diabetes risk score | baseline, 12 weeks, and 24 weeks
  change in diabetes risk score from baseline to 12 weeks and 24 weeks will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W True, MD, Principal Investigator — US Air Force
Locations (5):
- United States (5):
  - David Grant Medical Center, Travis AFB, California
  - Andrews Military Medical Center, Andrews Air Force Base Census Designated Place, Maryland
  - Nellis Family Medicine, Nellis Air Force Base, Nevada
  - Wright Patterson Medical Center, Wright-Patterson AFB, Ohio
  - Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas